CLINICAL TRIAL: NCT02882217
Title: Double-blind, Randomized, Dose-escalating, Placebo-controlled Study to Assess Pharmacokinetics, Safety, and Tolerability of XC-8 After Single and Multiple Oral Doses in Healthy Volunteers
Brief Title: Study to Assess Pharmacokinetics, Safety, and Tolerability of XC-8
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EURRUS Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PULM-XC8-03
Record Dates: First submitted 2016-08-01; First posted 2016-08-29 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Double-blind; Randomized; Dose-escalating; Placebo-controlled; Phase I; Healthy volunteers; Bronchial asthma; Histamine glutarimide; EURRUS
MeSH Terms: conditions — Asthma | interventions — histamine glutarimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- XC8 10mg (Active Comparator): Cohort 1: 8 subjects will be randomized in a 3:1 ratio to be treated either with 10mg XC8 (6 subjects) or placebo (2 subjects, see placebo arm)
  Interventions: Drug: XC8 (histamine glutarimide)
- XC8 50mg (Active Comparator): Cohort 2: 8 subjects will be randomized in a 3:1 ratio to be treated either with 50mg XC8 (6 subjects) or placebo (2 subjects, see placebo arm)
  Interventions: Drug: XC8 (histamine glutarimide)
- XC8 200mg (Active Comparator): Cohort 3: 16 subjects will be randomized in a 3:1 ratio to be treated either with 200mg XC8 (12 subjects) or placebo (4 subjects, see placebo arm)
  Interventions: Drug: XC8 (histamine glutarimide)
- Placebo (Placebo Comparator): Placebo comparator arm consists of 2 subjects in the cohorts 1 and 2 each and 4 subjects in the cohort 3.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC8 (histamine glutarimide)
  Arms: XC8 10mg; XC8 200mg; XC8 50mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study focusses on the evaluation of safety and tolerability of the XC8. The design of the study involves sequential dosing of cohorts (group of volunteers), taking increasing doses of the product after receiving conclusion and recommendation for further continuation of the study from the Dose Escalation Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 50 years;
2. Generally good health;
3. Body mass index of 19 to 30 kg/m² and >50 kg body weight;
4. Female subjects who are post-menopausal (no menstrual period for a minimum of 1 year), or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or practice a highly effective method of birth control, i.e. resulting in a failure rate of less than 1% per year when used consistently and correctly (e.g. implants, injectables, combined oral contraceptives, some intra-uterine devices, sexual abstinence, or vasectomized partner). The birth control method must have been applied for at least 1 cycle before and until 3 months after administration of the study medication.
5. Male subjects with a female partner of child-bearing potential agree to use a medically acceptable method of contraception (e.g. condoms, sexual abstinence, vasectomy) during the study, and until 3 months after the last intake of study medication.
6. Subjects are willing and able (in the opinion of the investigator) to understand and comply with the procedures and evaluations of the study.
7. Subjects must be willing and legally able to give written informed consent.

Exclusion Criteria:

1. Hepatic or renal disease; any other disease, which may influence the clinical trial results or may lead to health worsening during the trial (according to the investigator's opinion);
2. Clinically significant laboratory abnormalities;
3. Use of any medication, including prophylaxis, within 1 month before screening (including herbal preparations and nutritional supplements);
4. Positive test for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus HBV at Screening;
5. Irregular sleep (e.g. night work, sleep disturbances, insomnia, returning from another time zone, etc.);
6. History or current evidence of alcohol or drug abuse; alcohol or drug intake within 4 days before Screening;
7. History or current evidence of allergic reactions (including reactions to medications and food);
8. History or current evidence of symptomatic rhinitis within 2 years before Screening (allergic rhinitis, non-allergic rhinitis, or hay fever, excluding short-term viral infection - cold or influenza);
9. Blood or plasma donation, or surgery (in hospital) within 12 weeks of Screening;
10. Lactating or pregnant females; a positive pregnancy test before the first administration of investigational medicinal product or breastfeeding;
11. Current or previous (within 3 months of enrollment) treatment with another investigational drug and/or medical device or participation in another clinical study;
12. Previous enrollment in this clinical study;
13. Inability to understand or follow protocol instructions;
14. Smoking within 3 months before screening or throughout the study;
15. Lactose intolerance;
16. History of allergic reactions to XC-8 or any inactive ingredients of the trial medication;
17. Employees of the sponsor or subjects who are employees or relatives of the investigator;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events per treatment arm | Change from pre-dose up to Day 36
  Adverse events will be summarized descriptively by treatment arm. Verbatim terms will be mapped to preferred terms and organ systems using the current Medical Dictionary for Regulatory Activities version. For each preferred term, frequency counts and percentages will be calculated by cohort.The nature, severity, seriousness, and relationship to study medication will be summarized for all study subjects
Laboratory data | Changes from Day 1 (pre-dose) till Day 2
  Laboratory data (hematology, biochemistry and urinalysis) will be summarized by treatment arm. Changes from pre-dose will be presented using shift tables (employing the categories 'normal', 'abnormal, clinically not significant' and 'abnormal, clinically significant') and absolute changes in laboratory values, if appropriate.
Laboratory data | Changes from Day 8 (pre-dose) till Day 10
  Laboratory data (hematology, biochemistry and urinalysis) will be summarized by treatment arm. Changes from pre-dose will be presented using shift tables (employing the categories 'normal', 'abnormal, clinically not significant' and 'abnormal, clinically significant') and absolute changes in laboratory values, if appropriate.
Laboratory data | Changes from Day 8 (pre-dose) till Day 15
  Laboratory data (hematology, biochemistry and urinalysis) will be summarized by treatment arm. Changes from pre-dose will be presented using shift tables (employing the categories 'normal', 'abnormal, clinically not significant' and 'abnormal, clinically significant') and absolute changes in laboratory values, if appropriate.
Physical examination | Day 1
  Physical examination results will be listed for following: general appearance, skin, head, eyes, ears, nose, throat, neck (including thyroid), lymph nodes, chest, heart, abdomen (including liver examination), extremities, and nervous system.
Physical examination | Day 8
  Physical examination results will be listed for following: general appearance, skin, head, eyes, ears, nose, throat, neck (including thyroid), lymph nodes, chest, heart, abdomen (including liver examination), extremities, and nervous system.
12-lead ECG | Change from pre-dose till Day 2
  12-lead ECG results will be analyzed descriptively
12-lead ECG | Day 8
  12-lead ECG results will be analyzed descriptively
Vital signs | Changes from pre-dose till Day 36
  Vital signs (blood pressure, respiratory rate, pulse, and temperature) results will be analyzed descriptively.

SECONDARY OUTCOMES:
Pharmacokinetics of XC8 by assessing AUCinf | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4 and 8 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose); Day 8 to 11, 13 and 15 (Pre dose)
  Area under the plasma concentration-time curve extrapolated to infinity
Pharmacokinetics of XC8 by assessing Cmax | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4 and 8 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose); Day 8 to 11, 13 and 15 (Pre dose)
  Maximum plasma concentration
Pharmacokinetics of XC8 by assessing AUC0-tlast | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4 and 8 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose); Day 8 to 11, 13 and 15 (Pre dose)
  Area under the plasma concentration-time curve up to the last sampling time with a concentration above the limit of quantification
Pharmacokinetics of XC8 by assessing AUC0-24 | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4 and 8 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose); Day 8 to 11, 13 and 15 (Pre dose)
  Area under the plasma concentration-time curve up to 24 hours after study drug administration
Pharmacokinetics of XC8 by assessing t1/2 | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4 and 8 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose); Day 8 to 11, 13 and 15 (Pre dose)
  Terminal elimination half-life
Pharmacokinetics of XC8 by assessing Tmax | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4 and 8 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose); Day 8 to 11, 13 and 15 (Pre dose)
  Time to reach Cmax
Pharmacokinetics of XC8 by assessing λz | Day 1 and 21 (Pre dose, and 20 min, 40 min, 1, 2, 4 and 8 hours post dose), Day 2 and Day 22 (24 hours ±10 minutes post dose); Day 8 to 11, 13 and 15 (Pre dose)
  Apparent first order terminal elimination rate constant
Pharmacokinetics of XC8 by assessing Cav | Day 8 to 11, 13 and 15 (Pre dose); Day 21 (Pre dose, and 20 min, 40 min, 1, 2, 4 and 8 hours post dose), Day 22 (24 hours ±10 minutes post dose)
  Average concentration over one dosing interval
Pharmacodynamic analyses: blood eosinophils | changes from Day 1 (pre-dose) to Day 2 and Day 8 (pre-dose) to Day 22
Pharmacodynamic analyses: blood cytokines | changes from Day 1 (pre-dose) to Day 2 and Day 8 (pre-dose) to Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Schmutz, Mag.iur., Study Director — EURRUS Biotech GmbH
Locations (2):
- Karl Landsteiner Institut für experimentelle und klinische Pneumologie, Wolkersbergenstraße 1, Vienna, Austria
- Fraunhofer Institut für Toxikologie und Experimentelle Medizin ITEM, Feodor-Lynen-Str.15, Hanover, Germany

REFERENCES:
- [Derived] Renner A, Romanova J, Ferko B, Schmutz H, Nebolsin V, Muller M, Badorrek P, Marth K, Pohl W. Safety, pharmacokinetics and pharmacodynamics of a novel anti-asthmatic drug, XC8, in healthy probands. Pulm Pharmacol Ther. 2019 Dec;59:101852. doi: 10.1016/j.pupt.2019.101852. Epub 2019 Oct 6. PMID 31597083